CLINICAL TRIAL: NCT05244122
Title: Prevalence Effects in Visual Search: Theoretical and Practical Implications
Brief Title: PROJECT 2 EXAMPLE: Feedback X Prevalence Using Dermatology Stimuli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeremy M Wolfe, PhD, Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007P000646-A; R01EY017001 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Decision Making
Keywords: dermatology; signal detection theory; prevalence effects; base rate effects; online study; BESH
MeSH Terms: interventions — Prevalence

STUDY DESIGN:
Intervention Model Description: We tested ~800 observers on line in a study where they could participate in multiple conditions. We were looking for the effect of condition 1 on condition N+1
Masking Description: Observers were naive about the hypothesis but could have figured out if a specific condition did or did not have feedback, for example. Once the data were collected, investigators could determine what conditions were tested on which observers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feedback X Prevalence Using Dermatology Stimuli (Experimental): In this experiment, observers (Os) completed blocks of 80 trials. On each trial, they saw an image of a spot on the skin. They classified this as a melanoma (cancer) or a nevis (benign). Blocks could be of low prevalence (20% cancer cases, 16 images) or high prevalence (50%, 40 images). Os either did received trial by trial "Feedback" about their performance accuracy, or they did not. Thus, there were four types of block.
  Low prevalence, No Feedback Low prevalence, Feedback High prevalence, No Feedback High prevalence, Feedback Each of these four types of block was made available to Os on each of 6 days. Os could elect to view each of the four blocks each day. Our particular interest was in the effect of performing one block on performance on an immediately subsequent block.
  Interventions: Behavioral: Feedback; Behavioral: Prevalence

INTERVENTIONS:
Behavioral: Feedback — presence or absence of trial by trial feedback
Behavioral: Prevalence — In some blocks, skin cancer "target" images were present on 50% of trials (high prevalence). In other blocks, disease prevalence was 20%.

SUMMARY:
Imagine that a dermatologist spends the morning seeing patients who have been referred for suspicion of skin cancer. Many of them do, in fact, have skin lesions that require treatment. For this set of patients, disease 'prevalence' would be high. Suppose that the next task is to spend the afternoon giving annual screening exams to members of the general population. Here disease prevalence will be low. Would the morning's work influence decisions about patients in the afternoon? It is known from other contexts that recent history can influence current decisions and that target prevalence has an impact on decisions. In this study, decisions were decisions about skin lesions from individuals with varying degrees of expertise, using an online, medical imaging labelling app (DiagnosUs). This allowed examination of the effects of feedback history and prevalence in a single study. Blocks of trials could be of low or high prevalence, with or without feedback. Over 300,000 individual judgements were collected. (taken from Wolfe, J. M. (2022). How one block of trials influences the next: Persistent effects of disease prevalence and feedback on decisions about images of skin lesions in a large online study. . Cognitive Research: Principles and Implications (CRPI), 7, 10. doi: https://doi.org/10.1186/s41235-022-00362-0

DETAILED DESCRIPTION:
This description is based on a preregistration on the Open Science Framework site. Note that this is a "BESH" study. This type of research is not designed as a traditional clinical trial, but it is being reported here because of changes in NIH clinical trial reporting rules. This is one study from Project 2 of NE017001.

Levari et al (2018) found that people responded to a decrease in the prevalence of a stimulus by expanding their concept of it. Specifically, they asked observers to judge on each trial whether a dot, drawn from a blue-purple continuum, was blue or not. The results showed that observers were more likely to call ambiguous stimuli "blue" when blue items were less prevalent. In signal detection theory (SDT) terms, this is a liberal shift of response criterion. This is "prevalence induced concept change" (PICC). However, previous results obtained the opposite results in a long series of experiments on prevalence effects. The standard finding is that Os miss more targets at low prevalence. When blue is rare, they are less likely to call something blue. In SDT terms, this is a conservative criterion shift. This is the classic Low Prevalence Effect (LPE). In a round of earlier experiments, Lyu et al (2021) found that feedback is a critical variable. With trial-by-trial feedback, we get an LPE. With no feedback, the data usually show PICC results.

Do LPE and PICC effects show up when experts view stimuli in their expert domain? There is evidence for the LPE from search tasks (e.g. Evans, K. K., Birdwell, R. L., & Wolfe, J. M. (2013). If You Don't Find It Often, You Often Don't Find It: Why Some Cancers Are Missed in Breast Cancer Screening. . PLoS ONE 8(5): e64366. , 8(5), e64366. doi: doi:10.1371/journal.pone.0064366). However, PICC evidence has not been collected and there is no data from single item decision tasks like the "Is this dot blue?" task. This is important because criterion shifts of the sort described above can have obvious health care implications.

This study will repeat the basic "Is this dot blue" experiment using dermatology stimuli (Is this melanoma or just a nevus (a mole)?)

Hypotheses:

(H1) without feedback, Os are more likely to label a spot as cancer when cancer prevalence is low (prevalence-induced-concept-change).

(H2) that with feedback, Os are less likely to label a spot as cancer when cancer prevalence is low (classic low prevalence effect)

Dependent variable

The main dependent variable is the proportion of cancer responses as a function of the cancer prevalence in the image set, but we will also record reaction times.

Conditions

How many and which conditions will participants be assigned to?

Four conditions will be run, between observers.

1. 50% cancer images with feedback
2. 50% cancer images without feedback
3. 20% cancer images with feedback
4. 20% cancer images without feedback

Observers will make a simple 2-alternative forced-choice (2AFC) cancer/no cancer decision.

Observers will be awarded points based on the correctness of the answer (more correct, more points)

There will be 200 trials in each block. That will produce 40 target present trials in the low prevalence conditions which should produce a hit rate that is not too coarse.

Stimuli will be images of moles from the ISIC archive. Each image comes with a known answer of either melanoma (cancer) or nevus (negative).

Analyses

The data will produce a continuum from not-cancer to cancer based on the observers responses in the 50% with feedback condition. This will give yield a psychometric function rising (it may be assumed) from near 0% cancer responses to near 100%.

Using that ordering, psychometric functions will be generated for the other three conditions.

To examine the effect of prevalence and the presence and absence of feedback on observers' response behavior, \run a logistic regression with prevalence and feedback as factors in a generalized mixed model will be run using jamovi software.

The data will also be used to compute the signal detection measures of sensitivity (d') and criterion (c) based on the actual truth about the images. That is, "cancer" responses will be coded as True positives if the images show cancer and as "false positives" if they do not. T-tests will be performed to examine whether d' and/or c (criterion) change significantly as a function of prevalence and feedback.

Outliers and Exclusions

N/A

Sample Size

Separate blocks of trials will be run and conditions will be compared with unpaired t-tests.

G* Power says suggests 36 observers PER GROUP or a total of 144 observers for alpha = 0.05, power = 0.80. The plan will be to attempt to run 45 Os per group, anticipating about 20% loss of Os due to the vagaries of online testing.

ELIGIBILITY:
Inclusion Criteria:

* All welcome to enroll on line

Exclusion Criteria:

* Under 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1121 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Wolfe, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Visual Attention Lab, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD available on OSF. Other details available on request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available currently and indefinitely.
Access Criteria: OSF is publicly available. Other requests to jwolfe@bwh.harvard.edu

REFERENCES:
- [Result] Wolfe JM. How one block of trials influences the next: persistent effects of disease prevalence and feedback on decisions about images of skin lesions in a large online study. Cogn Res Princ Implic. 2022 Feb 2;7(1):10. doi: 10.1186/s41235-022-00362-0. PMID 35107667
- Available data/document: Individual Participant Data Set — https://osf.io/hck5n/ — This is the Open Science Framework page for these data. The title is Levari Exp. 17: Feedback X Prevalence using dermatology stimuli

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an online study. Participation was an option listed on the DiagnosUs site for 6 days in June, 2021.
Period: Overall Study
Arm/Group | Feedback X Prevalence Using Dermatology Stimuli
Started (This is the number of individuals who started the online study) | 1121
Completed a Full Block of Trials | 630 (Those 630 participants completed 2988 blocks in aggregate)
Completed (This is the number of participants who produced usable data. In an online study, participants often start a study but then decide they are not interested or don't have time. In any event, they do not complete the study.) | 803
Not Completed | 318
Not completed — Withdrawal by Subject | 318

BASELINE CHARACTERISTICS:
Arm/Group | Feedback X Prevalence Using Dermatology Stimuli
Number analyzed (Participants) | 803
Age, Customized [Count of Participants; unit: Participants]
  >=18 yrs | 803
Sex: Female, Male [Count of Participants; unit: Participants] — Population: sex data were not collected from any participants
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Expertise [Count of Participants; unit: Participants] — we have a crude categorization of expertise as shown below Medical Student 337 Pre-Med Student 174 No Medical Experience 145 Medical Doctor 54 Other Healthcare Professional 47 Nurse 25 Medical Technician 11 Physician Assistant 10
  Participants
    Medical Student | 337
    Pre-Med Student | 174
    No Medical Experience | 145
    Medical Doctor | 54
    Other Healthcare Professional | 47
    Nurse | 25
    Medical Technician | 11
    Physician Assistant | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in D' Between Pairs of Blocks.
Description: D' (d-prime) is defined as z-transform of the true positive rate - z-transform of false positive rate. True positive is when you say that a real melanoma is a melanoma. False positive is when you say that a nevis is a melanoma.
  A correction of 0.5 error is added to avoid calculation problems when z=0 or z=1.
  D' of zero indicates no ability to discriminate. D' > zero indicates some ability to discriminate.
  The change of interest is the D' for Block 2 when it follows Block 1 compared to the D' for Block 2 averaged across all conditions.
Time Frame: Participants could be in the study for as little as two blocks in one day up to 24 blocks collected over 6 days.
Population: Blocks having D' < 0.5 were excluded.
Measure: Mean (95% Confidence Interval); unit: z-score
Groups:
- Low Prevalence No Feedback First, Then Low Prevalence No Feedback; Low Prevalence No Feedback First, Then Low Prevalence With Feedback; Low Prevalence No Feedback First, Then High Prevalence No Feedback; Low Prevalence No Feedback First, Then High Prevalence With Feedback; Low Prevalence With Feedback First, Then Low Prevalence No Feedback; Low Prevalence With Feedback First, Then Low Prevalence With Feedback; Low Prevalence With Feedback First, Then High Prevalence No Feedback; Low Prevalence With Feedback First, Then High Prevalence With Feedback; High Prevalence No Feedback First, Then Low Prevalence No Feedback; High Prevalence No Feedback First, Then Low Prevalence With Feedback; High Prevalence No Feedback First, Then High Prevalence No Feedback; High Prevalence No Feedback First, Then High Prevalence With Feedback; High Prevalence With Feedback First, Then Low Prevalence No Feedback; High Prevalence With Feedback First, Then Low Prevalence With Feedback; High Prevalence With Feedback First, Then High Prevalence No Feedback; High Prevalence With Feedback First, Then High Prevalence With Feedback: Low prevalence means 20% (16 total) Melanoma images High prevalence means 50% (40 total) Melanoma images Feedback means participants were told if the response was correct after each trial.
  No Feedback means that they were not.
Arm/Group | Low Prevalence No Feedback First, Then Low Prevalence No Feedback | Low Prevalence No Feedback First, Then Low Prevalence With Feedback | Low Prevalence No Feedback First, Then High Prevalence No Feedback | Low Prevalence No Feedback First, Then High Prevalence With Feedback | Low Prevalence With Feedback First, Then Low Prevalence No Feedback | Low Prevalence With Feedback First, Then Low Prevalence With Feedback | Low Prevalence With Feedback First, Then High Prevalence No Feedback | Low Prevalence With Feedback First, Then High Prevalence With Feedback | High Prevalence No Feedback First, Then Low Prevalence No Feedback | High Prevalence No Feedback First, Then Low Prevalence With Feedback | High Prevalence No Feedback First, Then High Prevalence No Feedback | High Prevalence No Feedback First, Then High Prevalence With Feedback | High Prevalence With Feedback First, Then Low Prevalence No Feedback | High Prevalence With Feedback First, Then Low Prevalence With Feedback | High Prevalence With Feedback First, Then High Prevalence No Feedback | High Prevalence With Feedback First, Then High Prevalence With Feedback
Number analyzed (Participants) | 29 | 92 | 261 | 147 | 140 | 110 | 117 | 218 | 151 | 150 | 51 | 118 | 134 | 218 | 117 | 27
z-score | -0.138 [-0.335 to 0.0585] | .0754 [-0.126 to 0.277] | 0.023 [-0.0459 to 0.0920] | -.129 [-0.232 to -0.0259] | -0.0654 [-0.169 to 0.0382] | -0.139 [-0.259 to -0.0192] | 0.0603 [-0.0432 to 0.164] | 0.0582 [-0.0366 to 0.153] | 0.0792 [-0.0177 to 0.176] | 0.0452 [-0.0759 to 0.166] | -0.0123 [-0.168 to 0.143] | 0.035 [-0.0883 to 0.158] | 0.00902 [-0.107 to 0.125] | 0.00723 [-0.0947 to 0.109] | -0.106 [-0.202 to -0.0109] | 0.078 [-0.191 to 0.347]

2. Primary Outcome: Change in Criterion Between Pairs of Blocks.
Description: Criterion, c, corresponds to the position of the midpoint between the z-transformed probabilities of hits (correct yes responses) and false alarms (incorrect yes responses). It is calculated as -[z(p(h))+z(p(FA))]/2. The criterion, c, z-score quantifies the distance away from being unbiased in units of standard deviations. A Z-score of 0 is said to be unbiased. Negative values for c indicate a more relaxed criterion for saying yes. Positive numbers indicate a more strict criterion for saying yes.
Time Frame: Participants could be in the study for as little as two blocks in one day up to 24 blocks collected over 6 days.
Population: Blocks having D' < 0.5 were excluded.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Low Prevalence No Feedback First, Then Low Prevalence No Feedback | Low Prevalence No Feedback First, Then Low Prevalence With Feedback | Low Prevalence No Feedback First, Then High Prevalence No Feedback | Low Prevalence No Feedback First, Then High Prevalence With Feedback | Low Prevalence With Feedback First, Then Low Prevalence No Feedback | Low Prevalence With Feedback First, Then Low Prevalence With Feedback | Low Prevalence With Feedback First, Then High Prevalence No Feedback | Low Prevalence With Feedback First, Then High Prevalence With Feedback | High Prevalence No Feedback First, Then Low Prevalence No Feedback | High Prevalence No Feedback First, Then Low Prevalence With Feedback | High Prevalence No Feedback First, Then High Prevalence No Feedback | High Prevalence No Feedback First, Then High Prevalence With Feedback | High Prevalence With Feedback First, Then Low Prevalence No Feedback | High Prevalence With Feedback First, Then Low Prevalence With Feedback | High Prevalence With Feedback First, Then High Prevalence No Feedback | High Prevalence With Feedback First, Then High Prevalence With Feedback
Number analyzed (Participants) | 29 | 92 | 261 | 147 | 140 | 110 | 117 | 218 | 151 | 150 | 51 | 118 | 134 | 218 | 117 | 27
z-score | 0.0488 [-0.131 to 0.228] | 0.00147 [-0.0734 to 0.0763] | -0.026 [-0.0813 to 0.0293] | -0.0582 [-0.110 to -0.00631] | 0.182 [0.114 to 0.249] | 0.131 [0.0674 to 0.195] | 0.236 [0.166 to 0.305] | 0.0458 [0.0134 to 0.0783] | -0.0124 [-0.0752 to 0.0503] | 0.0136 [-0.0407 to 0.0678] | -0.00091 [-0.125 to 0.124] | 0.0186 [-0.0311 to 0.0683] | -0.187 [-0.276 to -0.0972] | -0.0762 [-0.119 to -0.0335] | -0.177 [-0.252 to -0.103] | -0.135 [-0.244 to -0.0260]

ADVERSE EVENTS:
Description: deaths and adverse events data were not collected in the minimal risk study
Arm/Group | Feedback X Prevalence Using Dermatology Stimuli
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Convenience sample of 803 participants is unbalanced. Online study lacks control over the display and ambient lighting. Other statistical analyses could be performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT05244122/Prot_SAP_000.pdf